CLINICAL TRIAL: NCT00644722
Title: Out-of-Hospital Intubation in Emergency Conditions With Either Metal Single Use or Reusable Laryngoscope Blades : Impact on Intubation Difficulties
Brief Title: Out-of-Hospital Intubation With Metal Single Use Laryngoscope Blades
Acronym: LAMETA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henri Mondor University Hospital (Other)
Collaborators: SFMU (Unknown)
Responsible Party: XAVIER COMBES MD, Service d'anesthésie reanimation SAMU 94 - CHU H MONDOR
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N° 2007-A00350-53
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Cardiac Arrest; Coma; Major Trauma; Respiratory Distress; Shock
Keywords: Intubation; Out-of-hospital; Laryngoscope; Blades; Emergency
MeSH Terms: conditions — Heart Arrest; Coma; Dyspnea; Shock; Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Single use metallic blades
  Interventions: Device: MacIntosh Green Lite (metal single use laryngoscope blades)
- 2 (Active Comparator): Classic reusable metallic blades
  Interventions: Device: MacIntosh Green Spec II (metal reusable laryngoscope blades)

INTERVENTIONS:
Device: MacIntosh Green Lite (metal single use laryngoscope blades) — metal single use laryngoscope blades
  Other Names: Truphatek company -Israel; Smiths Medical France company
  Arms: 1
Device: MacIntosh Green Spec II (metal reusable laryngoscope blades) — metal reusable laryngoscope blades
  Other Names: Truphatek company -Israel; Smiths Medical France company
  Arms: 2

SUMMARY:
New single use laryngoscope metal blades are available for intubation. This type of blade is safer than the reusable ones concerning the interhuman cross infection risk. No clinical studies have compared the two types of blades in the emergency context. The primary aim of this study is to demonstrate that single use blades are as efficient as the reusable ones concerning intubation conditions.

DETAILED DESCRIPTION:
All adult patients requiring tracheal intubation in the pre hospital emergency context will be included. All intubation will be performed by an emergency physician or a nurse specialized in anesthesia. For patients with spontaneous cardiac activity, rapid sequence intubation will be performed to allow intubation.

Comparisons studied will be : Intubation success rate at the first laryngoscopy, glottis exposure assessed by Cormack and Lehane classification, difficult intubation rate assessed by the Intubation Difficult Score (IDS), the need for alternative airway techniques and the immediate post intubation complications rate as vomiting, dental trauma, pulmonary inhalation, arterial desaturation , hypotension episodes and cardiac arrest occurrence.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients requiring out-of-hospital intubation

Exclusion Criteria:

* Patient under 18 years old
* Patients with criteria predictive of impossible intubation under direct laryngoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Intubation success rate during at the first laryngoscopy | 10 min

SECONDARY OUTCOMES:
glottis exposure assessed by Cormack and Lehane classification | 1 day
difficult intubation rate assessed by the Intubation Difficult Score (IDS) | 1 day
the need for alternative airway techniques and the immediate post intubation complications rate | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: XAVIER COMBES, MD, Principal Investigator — Service d'anesthésie reanimation SAMU 94 - CHU H MONDOR
Locations (1):
- Service d'anesthésie reanimation SAMU 94 - CHU H MONDOR - APHP, Créteil, Île-de-France Region, France